CLINICAL TRIAL: NCT01305486
Title: A Prospective, Multi-Center Study of Complex Ventral Hernia Repair Utilizing the XenMatrix™ Surgical Graft With Component Separation
Brief Title: A Study of Complex Ventral Hernia Repair Utilizing the XenMatrix™ Surgical Graft With Component Separation
Acronym: XenMatrix
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision, not safety related.
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: DVL-HE008
Record Dates: First submitted 2010-12-22; First posted 2011-02-28 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- XenMatrix

SUMMARY:
This will be an observational study designed to collect early, short- and long-term clinical outcomes of the XenMatrix™ Surgical Graft for complex ventral hernia repair. Subjects will be expected to attend follow up visits at 1, 6, 12, 18 and 24 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be able to undergo study procedures.
* Have signed an Informed Consent form (ICF).
* Be diagnosed with a ventral or incisional hernia that cannot be closed primarily in the opinion of the investigator.
* Requires a component separation repair with the use of a biological graft.

Exclusion Criteria:

* Subject is participating in another device or drug study.
* Subject has a life expectancy less than 4 years at the time of enrollment.
* Any condition in the opinion of the investigator that would preclude the use of the XenMatrix™ Surgical Graft, or preclude the subject from completing the follow-up requirements.
* Any subject with a defect the surgeon feels he/she cannot fully close.
* Subjects with a BMI > 50.
* Subjects with connective tissue disorders.
* Subjects with a history of cirrhosis.
* Subjects with renal failure requiring dialysis.
* Subjects on or suspected to be placed on chemotherapy or systemic immunosuppressive medications during any part of the study.
* Transplant recipients.
* Subjects taking corticosteroids for >6 months (pre or post surgery).
* Any bowel leak or infection that would preclude the use of the XenMatrix™ Surgical Graft in the opinion of the investigator.
* The subject lives approximately 2 hours away from the study site and compliance with follow up requirements will be difficult in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are diagnosed with a ventral or incisional hernia that require a component separation repair with the use of a biological graft.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To estimate the hernia recurrence rate of complex ventral hernias post repair with the XenMatrix™ Surgical Graft utilizing the component separation technique with several different tissue plane placements of the graft for up to 24 months post surgery. | 2 Years
  Any hernia which is identified or confirmed by the investigator in approximately the same position as the hernia repair during any follow up visit after a XenMatrix™ surgical graft has been placed will be considered a recurrent hernia.

SECONDARY OUTCOMES:
To assess perioperative, short-term and long-term complications in subjects with complex hernias repaired with XenMatrix™ Surgical Graft and component separation. | 2 Years
  Procedural and device related AEs collected from surgery until 24 months post surgery.
To assess the procedural time for XenMatrix™ Surgical Graft placement with component separation. | Day 0
  Procedure time will be defined as beginning when the investigator makes the initial skin incision and ending when the skin closure is completed (skin to skin).
To assess changes in subject quality of life (QOL) post repair with a XenMatrix™ Surgical Graft with component separation. | 2 years
  Changes in QOL will be assessed from baseline to 24 months utilizing the Short Form-36 (SF-36) version 2.
To assess clinical outcomes based on the tissue plane placement of the XenMatrix™ Surgical Graft. | 2 years
  Subjects who have their grafts placed in different tissue planes will have their recurrence rate, complication type and frequency examined to determine if there are any gross differences.

CONTACTS AND LOCATIONS:
Overall Officials: Karl LeBlanc, MD, Principal Investigator — Our Lady of the Lake Hospital
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States